CLINICAL TRIAL: NCT01410695
Title: A 24-week With Possible Extension, Prospective, Multicenter, Randomised, Double-blind, Controlled, 3-parallel Groups, Phase 2b/3 Study to Compare Efficacy and Safety of Masitinib at 3 and 6 mg/kg/Day to Methotrexate, With a Randomisation 1:1:1, in Treatment of Patients With Active Rheumatoid Arthritis With Inadequate Response to 1. Methotrexate or to 2. Any DMARD Including at Least One Biologic Drug if Patients Previously Failed Methotrexate or to 3. Methotrexate in Combination With Any DMARD Including Biologic Drugs
Brief Title: Masitinib in Refractory Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB06012
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; RA; masitinib; DMARD; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — masitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- masitinib 3 mg (Experimental): masitinib 3 mg/kg/day, tablets, orally, twice a day
  Interventions: Drug: masitinib 3 mg; Drug: Placebo (methotrexate)
- masitinib 6.0 mg (Experimental): masitinib 6.0 mg/kg/day, tablets, orally, twice a day
  Interventions: Drug: masitinib 6.0 mg; Drug: Placebo (methotrexate)
- methotrexate (Active Comparator): methotrexate at the dose of 15 or 20 mg per week
  Interventions: Drug: methotrexate; Drug: Placebo (masitinib)

INTERVENTIONS:
Drug: masitinib 3 mg
  Other Names: AB1010
  Arms: masitinib 3 mg
Drug: masitinib 6.0 mg
  Other Names: AB1010
  Arms: masitinib 6.0 mg
Drug: methotrexate
  Arms: methotrexate
Drug: Placebo (methotrexate)
  Arms: masitinib 3 mg; masitinib 6.0 mg
Drug: Placebo (masitinib)
  Arms: methotrexate

SUMMARY:
The objective is to compare efficacy and safety of masitinib at 3 and 6 mg/kg/day to methotrexate, with a randomisation 1:1:1, in treatment of patients with active rheumatoid arthritis with inadequate response to 1. methotrexate or to 2. any DMARD including at least one biologic drug if patients previously failed methotrexate or to 3. methotrexate in combination with any DMARD including biologic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with rheumatoid arthritis diagnosed according to American College of Rheumatology (ACR) criteria for at least 6 months
2. Patient with ACR functional class I-III
3. Patient who have active RA
4. Patient who failed (defined as active RA with stable dose during 3 months) methotrexate or any DMARD including biologics drugs if patients previously failed methotrexate or methotrexate in combination with any DMARD including biologics drugs
5. Patient with a disease onset at > 16 years of age

Exclusion Criteria:

1. Patient for whom the use of methotrexate is contraindicated as per its SPC
2. Patient with documented fibromyalgia
3. Patient with lactose intolerance
4. Patient presenting with cardiac disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
ACR50 | week 24

SECONDARY OUTCOMES:
ACR | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Tebib, MD, Principal Investigator — Centre Hospitalier Lyon Sud, Pierre-Bénite, France
Locations (1):
- ARTMEDI UPD s.r.o, Hostivice, Czechia